CLINICAL TRIAL: NCT00195663
Title: A Prospective Multi-Centre Randomised, Double-Blind, Active Comparator-Controlled, Parallel-Groups Study Comparing the Fully Human Monoclonal Anti-TNFα Antibody Adalimumab Given Every Second Week With Methotrexate Given Weekly and the Combination of Adalimumab and Methotrexate Administered Over 2 Years in Patients With Early Rheumatoid Arthritis (PREMIER).
Brief Title: Efficacy and Safety of Adalimumab and Methotrexate (MTX) Versus MTX Monotherapy in Subjects With Early Rheumatoid Arthritis
Acronym: PREMIER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DE013
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2010-02-25 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-06

CONDITIONS: Early Rheumatoid Arthritis
Keywords: Early Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adalimumab (Experimental): Participants received adalimumab 40 mg subcutaneous injection once every other week and placebo to methotrexate orally once a week during the 2-year double-blind treatment phase and then adalimumab 40 mg every other week for up to 8 years in the open-label extension.
  Interventions: Biological: Adalimumab; Drug: Methotrexate placebo
- Adalimumab + methotrexate (Experimental): Participants received adalimumab 40 mg subcutaneous injection once every other week and methotrexate orally once a week at a starting dose of 7.5 mg/week (could be escalated up to 20 mg/week) during the 2-year double-blind treatment phase. Participants received adalimumab 40 mg every other week for up to 8 years in the open-label extension phase.
  Interventions: Biological: Adalimumab; Drug: Methotrexate
- Methotrexate (Experimental): Participants received placebo to adalimumab subcutaneous injection once every other week and methotrexate orally once a week at a starting dose of 7.5 mg/week (could be escalated up to 20 mg/week) during the 2-year double-blind treatment phase. Participants received adalimumab 40 mg every other week for up to 8 years in the open-label extension phase.
  Interventions: Drug: Methotrexate; Biological: Adalimumab placebo

INTERVENTIONS:
Biological: Adalimumab
  Other Names: ABT-D2E7; Humira
  Arms: Adalimumab; Adalimumab + methotrexate
Drug: Methotrexate
  Arms: Adalimumab + methotrexate; Methotrexate
Biological: Adalimumab placebo
  Arms: Methotrexate
Drug: Methotrexate placebo
  Arms: Adalimumab

SUMMARY:
The purpose of the study is to assess the safety and efficacy of adalimumab in combination with methotrexate in patients with recent onset rheumatoid arthritis (RA), and to assess the long-term safety and maintenance of efficacy after treatment with adalimumab for up to 10 years.

DETAILED DESCRIPTION:
This study had an initial 2-year double-blind treatment period followed by an 8-year open-label extension period, for a total of up to 10 years study duration. The study was designed to assess the potential of adalimumab + methotrexate to improve signs and symptoms of disease and to inhibit radiographic progression in patients with recent onset (disease duration less than 3 years) rheumatoid arthritis not previously treated with methotrexate. Adalimumab is a human anti-tumor necrosis factor (TNF) monoclonal antibody.

ELIGIBILITY:
Inclusion Criteria:

* Subject was age 18 or older and in good health (Investigator discretion) with a recent stable medical history.
* Diagnosis of rheumatoid arthritis (RA) as defined by the 1987-revised American College of Rheumatology (ACR) criteria, with a disease duration less than 3 years, at least 8 swollen joints out of the 66 joints assessed, at least 10 tender joints out of the 68 joints assessed, at least 1 joint erosion or rheumatoid factor (RF) positivity, erythrocyte sedimentation rate (ESR) >= 28 mm/1h or C-reactive protein (CRP) >= 1.5 mg/dl

Exclusion Criteria:

* Chronic arthritis diagnosed before the age of 16
* Preceding treatment with MTX, cyclophosphamide, cyclosporin, azathioprine or more than 2 other disease-modifying anti-rheumatic drugs (DMARDs)
* Subject previously received anti-tumor necrosis factor (TNF) therapy
* Permanently wheelchair-bound or bedridden patients
* Subject considered by the investigator, for any reason, to be an unsuitable candidate for the study
* Female subject who is pregnant or breast-feeding or considering becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 799 (Actual)
Dates: Start 2000-12; Primary Completion 2004-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Carlson, Study Director — AbbVie
Locations (123):
- United States (31):
  - Site Reference ID/Investigator# 322, Scottsdale, Arizona
  - Site Ref # / Investigator 95957, La Jolla, California
  - Site Reference ID/Investigator# 429, La Jolla, California
  - Site Reference ID/Investigator# 2491, Los Angeles, California
  - Site Reference ID/Investigator# 2500, Denver, Colorado
  - Site Reference ID/Investigator# 762, Aventura, Florida
  - Site Reference ID/Investigator# 328, Sarasota, Florida
  - Site Reference ID/Investigator# 327, Tampa, Florida
  - Site Reference ID/Investigator# 325, Zephyrhills, Florida
  - Site Reference ID/Investigator# 302, Rockford, Illinois
  - Site Reference ID/Investigator# 319, Cumberland, Maryland
  - Site Ref # / Investigator 95960, Hagerstown, Maryland
  - Site Reference ID/Investigator# 326, Wheaton, Maryland
  - Site Reference ID/Investigator# 2533, Worcester, Massachusetts
  - Site Reference ID/Investigator# 336, Lincoln, Nebraska
  - Site Reference ID/Investigator# 318, Concord, New Hampshire
  - Site Reference ID/Investigator# 488, Durham, North Carolina
  - Site Reference ID/Investigator# 314, Dayton, Ohio
  - Site Reference ID/Investigator# 761, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 757, Eugene, Oregon
  - Site Reference ID/Investigator# 361, Lake Oswego, Oregon
  - Site Reference ID/Investigator# 316, Bethlehem, Pennsylvania
  - Site Reference ID/Investigator# 4649, Duncansville, Pennsylvania
  - Site Ref # / Investigator 96122, Austin, Texas
  - Site Reference ID/Investigator# 306, Austin, Texas
  - Site Reference ID/Investigator# 313, Austin, Texas
  - Site Reference ID/Investigator# 2437, Dallas, Texas
  - Site Reference ID/Investigator# 2532, Houston, Texas
  - Site Reference ID/Investigator# 758, Houston, Texas
  - Site Reference ID/Investigator# 321, Spokane, Washington
  - Site Reference ID/Investigator# 305, Yakima, Washington
- Australia (11):
  - Site Reference ID/Investigator# 310, Brisbane
  - Site Reference ID/Investigator# 755, Camperdown
  - Site Reference ID/Investigator# 337, Clayton
  - Site Reference ID/Investigator# 331, Darlinghurst, Sydney
  - Site Reference ID/Investigator# 745, Kogarah
  - Site Reference ID/Investigator# 738, Maroochydore
  - Site Reference ID/Investigator# 335, New Lambton
  - Site Reference ID/Investigator# 737, Shenton Park
  - Site Reference ID/Investigator# 307, South Hobart
  - Site Reference ID/Investigator# 427, West Heidelberg
  - Site Reference ID/Investigator# 739, Woodville
- Site Reference ID/Investigator# 344, Vienna, Austria
- Belgium (7):
  - Site Reference ID/Investigator# 753, Brussels
  - Site Reference ID/Investigator# 308, Brussels
  - Site Reference ID/Investigator# 752, Brussels
  - Site Reference ID/Investigator# 748, Diepenbeek
  - Site Reference ID/Investigator# 6136, Ghent
  - Site Ref # / Investigator 98256, Leuven
  - Site Reference ID/Investigator# 333, Liège
- Canada (14):
  - Site Ref # / Investigator 98199, North York, Ontario
  - Site Reference ID/Investigator# 4646, Edmonton
  - Site Reference ID/Investigator# 303, Hamilton
  - Site Reference ID/Investigator# 330, Hamilton
  - Site Reference ID/Investigator# 4634, Montreal
  - Site Reference ID/Investigator# 311, Montreal
  - Site Reference ID/Investigator# 309, Newmarket
  - Site Reference ID/Investigator# 304, Pointe-Claire
  - Site Reference ID/Investigator# 4633, Richmond
  - Site Reference ID/Investigator# 763, St. John's
  - Site Reference ID/Investigator# 4635, Toronto
  - Site Reference ID/Investigator# 490, Toronto
  - Site Reference ID/Investigator# 760, Victoria
  - Site Reference ID/Investigator# 4632, Winnipeg
- Czechia (3):
  - Site Reference ID/Investigator# 754, Hradec Králové
  - Site Reference ID/Investigator# 332, Pilsen
  - Site Reference ID/Investigator# 734, Prague
- Site Ref # / Investigator 95878, Gråsten, Denmark
- Finland (2):
  - Site Reference ID/Investigator# 6135, Heinola
  - Site Ref # / Investigator 6134, Helsinki
- France (6):
  - Site Reference ID/Investigator# 428, Bobigny
  - Site Reference ID/Investigator# 348, Montpellier
  - Site Reference ID/Investigator# 4650, Paris
  - Site Reference ID/Investigator# 3415, Pierre-Bénite
  - Site Reference ID/Investigator# 733, Rennes
  - Site Reference ID/Investigator# 346, Strasbourg
- Germany (11):
  - Site Reference ID/Investigator# 4631, Berlin
  - Site Reference ID/Investigator# 759, Berlin
  - Site Reference ID/Investigator# 3417, Buch
  - Site Reference ID/Investigator# 4630, Erlangen
  - Site Reference ID/Investigator# 347, Freiburg im Breisgau
  - Site Reference ID/Investigator# 742, Görlitz
  - Site Reference ID/Investigator# 746, Leipzig
  - Site Ref # / Investigator 98125, Munich
  - Site Reference ID/Investigator# 339, Munich
  - Site Reference ID/Investigator# 744, Ratingen
  - Site Reference ID/Investigator# 338, Vogelsang-Gommern
- Ireland (2):
  - Site Reference ID/Investigator# 740, Cork
  - Site Reference ID/Investigator# 751, Dublin
- Italy (4):
  - Site Ref # / Investigator 95719, Genoa
  - Site Reference ID/Investigator# 323, Naples
  - Site Reference ID/Investigator# 345, Udine
  - Site Reference ID/Investigator# 756, Verona
- Netherlands (4):
  - Site Reference ID/Investigator# 343, Groningen
  - Site Reference ID/Investigator# 6133, Leiden
  - Site Reference ID/Investigator# 317, Maastricht
  - Site Reference ID/Investigator# 315, Nijmegen
- Norway (2):
  - Site Ref # / Investigator 95800, Oslo
  - Site Ref # / Investigator 95875, Oslo
- Site Reference ID/Investigator# 3426, Piešťany, Slovakia
- Spain (9):
  - Site Ref # / Investigator 96121, Alicante
  - Site Reference ID/Investigator# 735, Alicante
  - Site Reference ID/Investigator# 1525, Barcelona
  - Site Reference ID/Investigator# 1528, Barcelona
  - Site Reference ID/Investigator# 750, Guadalajara
  - Site Reference ID/Investigator# 1526, Madrid
  - Site Reference ID/Investigator# 741, Madrid
  - Site Reference ID/Investigator# 390, Santiago de Compostela
  - Site Reference ID/Investigator# 749, Seville
- Sweden (7):
  - Site Reference ID/Investigator# 728, Stockholm
  - Site Reference ID/Investigator# 2565, Stockholm
  - Site Reference ID/Investigator# 4638, Stockholm
  - Site Ref # / Investigator 96126, Umeå
  - Site Reference ID/Investigator# 747, Uppsala
  - Site Ref # / Investigator 96120, Västerås
  - Site Reference ID/Investigator# 736, Västerås
- Site Reference ID/Investigator# 334, Lausanne, Switzerland
- United Kingdom (6):
  - Site Ref # / Investigator 96116, Bangor
  - Site Ref # / Investigator 95877, Cambridge
  - Site Ref # / Investigator 98258, Hereford
  - Site Ref # / Investigator 95795, Leeds
  - Site Ref # / Investigator 95958, London
  - Site Ref # / Investigator 98255, Newcastle upon Tyne

REFERENCES:
- [Derived] Smolen J, Fleischmann R, Aletaha D, Li Y, Zhou Y, Sainsbury I, Galindo IL. Disease activity improvements with optimal discriminatory ability between treatment arms: applicability in early and established rheumatoid arthritis clinical trials. Arthritis Res Ther. 2019 Nov 10;21(1):231. doi: 10.1186/s13075-019-2005-9. PMID 31707982
- [Derived] Smolen JS, van Vollenhoven RF, Florentinus S, Chen S, Suboticki JL, Kavanaugh A. Predictors of disease activity and structural progression after treatment with adalimumab plus methotrexate or continued methotrexate monotherapy in patients with early rheumatoid arthritis and suboptimal response to methotrexate. Ann Rheum Dis. 2018 Nov;77(11):1566-1572. doi: 10.1136/annrheumdis-2018-213502. Epub 2018 Aug 3. PMID 30076156
- [Derived] Keystone EC, Breedveld FC, Kupper H, Li Y, Florentinus S, Sainsbury I. Long-term use of adalimumab as monotherapy after attainment of low disease activity with adalimumab plus methotrexate in patients with rheumatoid arthritis. RMD Open. 2018 Jun 13;4(1):e000637. doi: 10.1136/rmdopen-2017-000637. eCollection 2018. PMID 29955381
- [Derived] Keystone EC, Breedveld FC, van der Heijde D, van Vollenhoven RF, Emery P, Smolen JS, Sainsbury I, Florentinus S, Kupper H, Chen K, Kavanaugh A. Achieving comprehensive disease control in patients with early and established rheumatoid arthritis treated with adalimumab plus methotrexate versus methotrexate alone. RMD Open. 2017 Sep 26;3(2):e000445. doi: 10.1136/rmdopen-2017-000445. eCollection 2017. PMID 29018564
- [Derived] Moller B, Everts-Graber J, Florentinus S, Li Y, Kupper H, Finckh A. Low Hemoglobin and Radiographic Damage Progression in Early Rheumatoid Arthritis: Secondary Analysis From a Phase III Trial. Arthritis Care Res (Hoboken). 2018 Jun;70(6):861-868. doi: 10.1002/acr.23427. Epub 2018 Apr 25. PMID 28950430
- [Derived] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778
- [Derived] Landewe R, Smolen JS, Florentinus S, Chen S, Guerette B, van der Heijde D. Existing joint erosions increase the risk of joint space narrowing independently of clinical synovitis in patients with early rheumatoid arthritis. Arthritis Res Ther. 2015 May 21;17(1):133. doi: 10.1186/s13075-015-0626-1. PMID 25994819
- [Derived] Landewe R, Ostergaard M, Keystone EC, Florentinus S, Liu S, van der Heijde D. Analysis of integrated radiographic data from two long-term, open-label extension studies of adalimumab for the treatment of rheumatoid arthritis. Arthritis Care Res (Hoboken). 2015 Feb;67(2):180-6. doi: 10.1002/acr.22426. PMID 25073879
- [Derived] Keystone EC, Haraoui B, Guerette B, Mozaffarian N, Liu S, Kavanaugh A. Clinical, functional, and radiographic implications of time to treatment response in patients with early rheumatoid arthritis: a posthoc analysis of the PREMIER study. J Rheumatol. 2014 Feb;41(2):235-43. doi: 10.3899/jrheum.121468. Epub 2013 Dec 1. PMID 24293583
- [Derived] Keystone EC, Breedveld FC, van der Heijde D, Landewe R, Florentinus S, Arulmani U, Liu S, Kupper H, Kavanaugh A. Longterm effect of delaying combination therapy with tumor necrosis factor inhibitor in patients with aggressive early rheumatoid arthritis: 10-year efficacy and safety of adalimumab from the randomized controlled PREMIER trial with open-label extension. J Rheumatol. 2014 Jan;41(1):5-14. doi: 10.3899/jrheum.130543. Epub 2013 Nov 15. PMID 24241487
- [Derived] Smolen JS, van der Heijde DM, Keystone EC, van Vollenhoven RF, Goldring MB, Guerette B, Cifaldi MA, Chen N, Liu S, Landewe RB. Association of joint space narrowing with impairment of physical function and work ability in patients with early rheumatoid arthritis: protection beyond disease control by adalimumab plus methotrexate. Ann Rheum Dis. 2013 Jul;72(7):1156-62. doi: 10.1136/annrheumdis-2012-201620. Epub 2012 Aug 22. PMID 22915617
- [Derived] Strand V, Rentz AM, Cifaldi MA, Chen N, Roy S, Revicki D. Health-related quality of life outcomes of adalimumab for patients with early rheumatoid arthritis: results from a randomized multicenter study. J Rheumatol. 2012 Jan;39(1):63-72. doi: 10.3899/jrheum.101161. Epub 2011 Nov 1. PMID 22045836
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 94 sites in 15 countries between January 2001 and April 2004.
Pre-assignment Details: Patients who had been receiving a previous disease-modifying anti-rheumatic drug (DMARD) participated in a 4-week washout period during which the DMARD was withdrawn. Otherwise, there was a one-week washout period after the Screening visit.
Period: 2-year Double-blind Treatment Period
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Started | 257 | 274 | 268
Completed | 164 | 166 | 196
Not Completed | 93 | 108 | 72
Not completed — Adverse Event | 21 | 27 | 32
Not completed — Death | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 15 | 18 | 12
Not completed — Lack of Efficacy | 47 | 52 | 13
Not completed — Protocol Violation | 6 | 6 | 4
Not completed — Planned selection criteria | 0 | 1 | 0
Not completed — Recovery | 1 | 0 | 1
Not completed — Administrative reasons | 3 | 2 | 9
Period: Open-Label Extension Period
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Started | 155 | 159 | 183
Completed | 79 | 85 | 86
Not Completed | 76 | 74 | 97
Not completed — Adverse Event | 21 | 32 | 36
Not completed — Lost to Follow-up | 9 | 2 | 6
Not completed — Recovery | 0 | 2 | 2
Not completed — Protocol Violation | 3 | 4 | 4
Not completed — Death | 2 | 2 | 2
Not completed — Withdrawal by Subject | 16 | 15 | 22
Not completed — Lack of Efficacy | 14 | 6 | 12
Not completed — Administrative reasons | 11 | 11 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate | Total
Number analyzed (Participants) | 257 | 274 | 268 | 799
Age Continuous [Mean (Standard Deviation); unit: years] | 52.0 (13.1) | 52.1 (13.5) | 51.9 (14.0) | 52.0 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 212 | 193 | 595
  Male | 67 | 62 | 75 | 204

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Meeting American College of Rheumatology 50% (ACR50) Response Criteria at Week 52
Description: American College of Rheumatology 50% (ACR50) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 50% improvement in tender joint count;
  * ≥ 50% improvement in swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI));
    * Acute phase reactant value (C-Reactive Protein).
  Participants who withdrew early were considered non-responders.
Time Frame: Baseline and 52 Weeks
Population: The Full Analysis Set consisted of all patients who were randomized and who received at least one dose of double-blinded study medication. Participants with insufficient data to calculate ACR50 at Week 52 or who withdrew early were considered non-responders.
Measure: Number; unit: participants
Groups:
- Methotrexate: Participants received placebo to adalimumab subcutaneous injection once every other week and methotrexate orally once a week at a starting dose of 7.5 mg/week (could be escalated up to 20 mg/week) during the 2-year double-blind treatment phase.
- Adalimumab: Participants received adalimumab 40 mg subcutaneous injection once every other week and placebo to methotrexate orally once a week during the 2-year double-blind treatment phase.
- Adalimumab + Methotrexate: Participants received adalimumab 40 mg subcutaneous injection once every other week and methotrexate orally once a week at a starting dose of 7.5 mg/week (could be escalated up to 20 mg/week) during the 2-year double-blind treatment phase.
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
participants | 118 | 113 | 165
Statistical Analysis 1: Comparison: Methotrexate vs Adalimumab + Methotrexate; The study was powered to demonstrate the superiority of adalimumab + MTX combination therapy vs. MTX monotherapy in the proportion of subjects who achieved an ACR50 response at 52 weeks. Power calculations were based on 250 subjects in each group using a chi-squared test with a continuity correction and an alpha = 0.05 significance level. With 250 subjects in each group, a difference of 0.13 in response rates could be detected with 80% power; Test type: Superiority or Other; p < 0.001, Chi-squared, Corrected — Statistical tests were performed in a hierarchical manner. If there was a statistically significant difference in favor of adalimumab + MTX combination treatment, the second primary analysis of the modified Total Sharp Score was to be performed

2. Primary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) at Week 52
Description: The modified Total Sharp Score (mTSS) is a measure of change in joint health. Digitized images of radiographs of hands and feet obtained at screening and Week 52 were scored in a blinded manner. Joints were scored for erosions on a scale from 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale from 0 (no damage) to 4 (ankylosis or complete dislocation). Erosion scores and narrowing scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]). An increase in mTSS from Baseline represents disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease represents improvement.
Time Frame: Baseline and Week 52
Population: Full analysis set. For participants with missing data, mTSS was imputed by linear extrapolation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
units on a scale | 5.7 (12.7) [-58.0 to 78.5] | 3.0 (11.2) | 1.3 (6.5) [-68.0 to 29.5]
Statistical Analysis 1: Comparison: Methotrexate vs Adalimumab + Methotrexate; Statistical tests were performed in a hierarchical manner. If there was a statistically significant difference in favor of adalimumab + MTX combination treatment on the ACR50 response, the second primary analysis of modified TSS would be performed; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire - Disability Index (HAQ-DI) at Week 52
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Negative mean changes from Baseline in the overall score indicate improvement.
Time Frame: Baseline and Week 52
Population: Full analysis set with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 191 | 191 | 213
units on a scale | -0.8 (0.6) | -0.8 (0.7) | -1.1 (0.6)
Statistical Analysis 1: Comparison: Methotrexate vs Adalimumab + Methotrexate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Participants Meeting American College of Rheumatology 50% (ACR50) Response Criteria at Week 104
Description: American College of Rheumatology 50% (ACR50) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 50% improvement in tender joint count;
  * ≥ 50% improvement in swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * Acute phase reactant value (C-Reactive Protein).
  Participants withdrawing early were considered non-responders.
Time Frame: Baseline and Week 104
Population: Full analysis set. Participants with insufficient data to calculate ACR50 at Week 104 or who withdrew early were considered non-responders.
Measure: Number; unit: participants
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
participants | 110 | 101 | 158
Statistical Analysis 1: Comparison: Methotrexate vs Adalimumab + Methotrexate; Test type: Superiority or Other; p < 0.001, Chi-squared

5. Secondary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) at Week 104
Description: The modified Total Sharp Score (mTSS) is a measure of change in joint health. Digitized images of radiographs of hands and feet obtained at screening and Week 104 were scored in a blinded manner. Joints were scored for erosions on a scale of 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale of 0 (no damage) to 4 (ankylosis or complete dislocation). Erosion scores and narrowing scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]). An increase in mTSS from Baseline represents disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease represents improvement.
Time Frame: Baseline and Week 104
Population: Full analysis set. For participants with missing data, mTSS was imputed by linear extrapolation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
units on a scale | 10.4 (21.7) | 5.5 (15.8) | 1.9 (8.3)
Statistical Analysis 1: Comparison: Methotrexate vs Adalimumab + Methotrexate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Participants Who Achieved Clinical Remission, Defined as a Disease Activity 28 (DAS28) Score < 2.6 at Week 52
Description: The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C reactive protein, and general health were included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
Time Frame: Week 52
Population: Full analysis set. Participants with insufficient data to calculate DAS28 at Week 52 or who withdrew early were considered non-responders.
Measure: Number; unit: participants
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
participants | 53 | 64 | 115
Statistical Analysis 1: Comparison: Methotrexate vs Adalimumab + Methotrexate; Test type: Superiority or Other; p < 0.001, Chi-squared

7. Secondary Outcome: Change From Baseline in the Physical Component of the Short Form-36 Health Status Survey (SF-36) at Week 52
Description: The SF-36 determined participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 comprise the physical component of the SF-36. Scores on each item were summed and averaged (range = 0-100); increases from Baseline indicate improvement.
Time Frame: Baseline and Week 52
Population: Full analysis set with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 181 | 181 | 198
units on a scale | 12.5 (9.6) | 12.6 (10.0) | 16.7 (10.2)
Statistical Analysis 1: Comparison: Methotrexate vs Adalimumab + Methotrexate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Number of Participants With Major Clinical Response After 104 Weeks of Treatment
Description: Major clinical response was defined as an American College of Rheumatology 70% (ACR70) response for any six continuous months, over 104 weeks of treatment. A participant was a responder if the following criteria for improvement from Baseline were met:
  * ≥ 70% improvement in tender joint count;
  * ≥ 70% improvement in swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * Acute phase reactant value (C-Reactive Protein).
  Participants withdrawing early were non-responders.
Time Frame: Any 6 continuous months from Baseline to Week 104
Population: Full analysis set.
Measure: Number; unit: participants
Groups:
- Methotrexate Weekly: Participants received placebo to adalimumab subcutaneous injection once every other week and methotrexate orally once a week at a starting dose of 7.5 mg/week (could be escalated up to 20 mg/week) during the 2-year double-blind treatment phase.
Arm/Group | Methotrexate Weekly | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
participants | 70 | 67 | 130
Statistical Analysis 1: Comparison: Methotrexate Weekly vs Adalimumab + Methotrexate; Test type: Superiority or Other; p < 0.001, Chi-squared

9. Secondary Outcome: Change From Baseline in the Mental Component of the Short Form-36 Health Status Survey (SF-36) at Week 52
Description: The SF-36 determined participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 5-8 comprise the mental component of the SF-36. Scores on each item were summed and averaged (range = 0-100); increases from Baseline indicate improvement.
Time Frame: Baseline and Week 52
Population: Full analysis set with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 181 | 181 | 198
units on a scale | 6.5 (11.0) | 7.1 (12.3) | 7.2 (13.1)
Statistical Analysis 1: Comparison: Methotrexate vs Adalimumab + Methotrexate; Test type: Superiority or Other; p = 0.5402, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Number of Participants Meeting American College of Rheumatology 50% (ACR50) Response Criteria at Weeks 26 and 76
Description: as for outcome 4
Time Frame: Baseline and Weeks 26 and 76
Population: Full analysis set. Participants with insufficient data to calculate ACR50 or who withdrew early were considered non-responders.
Measure: Number; unit: participants
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
participants
  Week 26 | 104 | 96 | 157
  Week 76 | 114 | 114 | 161

11. Secondary Outcome: Number of Participants Meeting American College of Rheumatology 20% (ACR20) Response Criteria During the Double-blind Phase
Description: American College of Rheumatology 20% (ACR20) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 20% improvement in tender joint count;
  * ≥ 20% improvement in swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * Acute phase reactant value (C-Reactive Protein).
  Participants withdrawing early were considered non-responders.
Time Frame: Baseline and Weeks 26, 52, 76, and 104
Population: Full analysis set. Participants with insufficient data to calculate ACR20 or who withdrew early were considered non-responders.
Measure: Number; unit: participants
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
participants
  Week 26 | 158 | 146 | 184
  Week 52 | 161 | 149 | 195
  Week 76 | 154 | 137 | 185
  Week 104 | 144 | 135 | 186

12. Secondary Outcome: Number of Participants Meeting American College of Rheumatology 70% (ACR70) Response Criteria During the Double-blind Phase
Description: American College of Rheumatology 70% (ACR70) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 70% improvement in tender joint count;
  * ≥ 70% improvement in swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire Disability Index [HAQ-DI]);
    * Acute phase reactant value (C-Reactive Protein).
  Participants withdrawing early were considered non-responders.
Time Frame: Baseline and Weeks 26, 52, 76, and 104
Population: Full analysis set. Participants with insufficient data to calculate ACR70 or who withdrew early were considered non-responders.
Measure: Number; unit: participants
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
participants
  Week 26 | 57 | 54 | 114
  Week 52 | 70 | 71 | 122
  Week 76 | 75 | 79 | 127
  Week 104 | 73 | 77 | 125

13. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire - Disability Index (HAQ-DI) During the Double-blind Treatment Phase
Description: as for outcome 3
Time Frame: Baseline and Weeks 12, 26, 76, and 104
Population: Full analysis set with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
units on a scale
  Week 12 [N=236, 246, 252] | -0.6 (0.6) | -0.6 (0.6) | -0.8 (0.6)
  Week 26 [N=217, 222, 240] | -0.8 (0.6) | -0.8 (0.7) | -0.9 (0.6)
  Week 76 [N= 176, 175, 207] | -0.8 (0.6) | -0.9 (0.7) | -1.0 (0.7)
  Week 104 [166, 162, 201] | -0.9 (0.6) | -0.9 (0.6) | -1.0 (0.7)

14. Secondary Outcome: Number of Participants With Improvement in the HAQ-DI Score ≥ 0.3 During the Double-blind Treatment Phase
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability.
Time Frame: Baseline and Weeks 26, 52, 76, and 104
Population: Full analysis set. Missing values were considered to be < 0.3.
Measure: Number; unit: participants
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
participants
  Week 26 | 172 | 169 | 200
  Week 52 | 158 | 151 | 186
  Week 76 | 144 | 145 | 173
  Week 104 | 137 | 132 | 171

15. Secondary Outcome: Change From Baseline in Health Utilities Index Mark 2 and Mark 3 (HUI 2/3) During the Double-blind Treatment Phase
Description: The HUI 2/3 is an assessment of various aspects of participants' health and ability to perform various tasks on a day-to-day basis, including reading, seeing, hearing, speaking, general outlook on life, pain/discomfort, ability to walk, use of hands, memory, ability to think/solve, and ability to perform basic activities such as eating, bathing, and dressing. The HUI 2/3 is a combined 15-item questionnaire based on a recall period of the previous 4 weeks. HUI-2 and HUI-3 scores are calculated independently. The HUI-2 score includes 6 attributes: Sensation, Mobility, Emotion, Cognition, Self-Care, and Pain. The HUI-3 score is comprised of 8 attributes: Vision, Hearing, Speech, Ambulation, Dexterity, Emotion, Cognition, and Pain.
  The range of each score is from 0 (dead) to 1 (perfect health). An increase from Baseline indicates improvement.
Time Frame: Baseline and Weeks 26, 52, and 104
Population: Full analysis set with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
units on a scale
  HUI-2: Week 26 [N=192, 187, 205] | 0.2 (0.2) | 0.2 (0.2) | 0.2 (0.2)
  HUI-2: Week 52 [N=179, 162, 189] | 0.2 (0.2) | 0.2 (0.2) | 0.2 (0.2)
  HUI-2: Week 104 [N=152, 136, 174] | 0.2 (0.2) | 0.2 (0.2) | 0.2 (0.2)
  HUI-3: Week 26 [N=192, 189, 205] | 0.3 (0.3) | 0.3 (0.3) | 0.3 (0.3)
  HUI-3: Week 52 [N=177, 164, 190] | 0.3 (0.3) | 0.3 (0.3) | 0.4 (0.3)
  HUI-3: Week 104 [N=154, 138, 177] | 0.3 (0.2) | 0.4 (0.3) | 0.4 (0.3)

16. Secondary Outcome: Change From Baseline in the Short Form-36 Health Status Survey (SF-36) During the Double-blind Treatment Phase
Description: The SF-36 determined participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 comprise the physical component and items 5-8 comprise the mental component of the SF-36. Scores on each item were summed and averaged (range = 0-100); increases from Baseline indicate improvement.
Time Frame: Baseline and Weeks 26 and 104
Population: Full analysis set with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
units on a scale
  Physical Component: Week 26 [N=199, 204, 221] | 11.2 (10.0) | 10.8 (10.2) | 14.7 (10.2)
  Physical Component: Week 104 [160, 157, 189] | 12.4 (10.3) | 13.4 (9.7) | 16.8 (11.2)
  Mental Component: Week 26 [N=199, 204, 221] | 7.0 (11.6) | 5.2 (13.5) | 6.3 (12.1)
  Mental Component: Week 104 [N=160, 157, 189] | 8.1 (10.9) | 6.6 (13.5) | 6.8 (12.0)

17. Secondary Outcome: Numeric American College of Rheumatology (ACR-N) During the Double-blind Treatment Phase
Description: ACR-N is a composite, continuous variable which measures the percentage of improvement from Baseline in individual participants based on the 7 core set variables of the ACR. ACR-N is defined as the smallest percent change from Baseline of 3 measures: tender joint counts (TJC), swollen joint counts (SJC), and the median percent improvement in the 5 remaining measures (Patient's Assessment of Pain, Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity, Health Assessment Questionnaire - Disability Index [HAQ-DI], and C-Reactive Protein). A positive ACR-N value indicates improvement; a negative ACR-N value indicates worsening; ACR-N of 0 indicates no change.
Time Frame: Baseline and Weeks 26, 52, 76, and 104
Population: Full analysis set with available data.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
percent change
  Week 26 [N=218, 224, 244] | 44.7 (42.2) | 39.1 (43.3) | 57.0 (42.2)
  Week 52 [N=194, 193, 220] | 50.2 (48.2) | 44.4 (52.2) | 66.3 (34.8)
  Week 76 [N=181, 179, 211] | 56.1 (38.1) | 51.5 (56.8) | 68.8 (31.3)
  Week 104 [N=168, 167, 203] | 57.3 (37.1) | 54.0 (42.7) | 71.4 (31.0)

18. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS28) During the Double-blind Treatment Phase
Description: The DAS28 is a composite score of rheumatoid arthritis disease activity derived from the following variables:
  * 28 tender joint counts,
  * 28 swollen joint counts,
  * C-reactive protein, and
  * Patient's global assessment of disease activity.
  Scores on the DAS28 range from 0 to 10. A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Baseline and Weeks 26, 52, 76, and 104
Population: Full analysis set with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
units on a scale
  Week 26 [N=209, 218, 229] | -2.6 (1.3) | -2.4 (1.4) | -3.2 (1.3)
  Week 52 [N=184, 185, 206] | -2.8 (1.4) | -2.8 (1.5) | -3.6 (1.3)
  Week 76 [N=173, 173, 197] | -3.1 (1.2) | -3.0 (1.5) | -3.7 (1.3)
  Week 104 [N=161, 158, 191] | -3.1 (1.4) | -3.2 (1.4) | -3.8 (1.3)

19. Secondary Outcome: Change From Baseline in Joint Erosion Score During the Double-blind Treatment Period
Description: Digitized images of radiographs of hands and feet obtained at screening and during the study were scored in a blinded manner. Joints on each hand/wrist (17 joints) and each forefoot (6 joints) were scored for erosions on a scale of 0 = no erosions; 1 = 1 discrete erosion or ≤20% joint involvement; 2 = 2 separate quadrants with erosion or 21-40% joint involvement; 3 = 3 separate quadrants with erosion or 41-60% joint involvement; 4 = all 4 quadrants with erosion or 61-80% joint involvement; and 5 = extensive destruction with >80% joint involvement. Scores were summed to calculate the total erosion score, which ranges from 0 (no erosion)to 230 (worst). A large increase in erosion score is indicative of worsening, whereas a small change or no change is indicative of inhibition of joint erosion.
Time Frame: Baseline and Weeks 52 and 104
Population: Full analysis set. Missing values were imputed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
units on a scale
  Week 52 | 3.7 (8.4) | 1.7 (5.7) | 0.8 (3.3)
  Week 104 | 6.4 (14.3) | 3.0 (8.3) | 1.0 (4.7)

20. Secondary Outcome: Change From Baseline in Joint Space Narrowing Score During the Double-blind Treatment Period
Description: Digitized images of radiographs of hands and feet obtained at screening and during the study were scored in a blinded manner. Joint space narrowing (JSN) scores were recorded for each hand/wrist (16 joints) and each forefoot (5 joints) on a 5-point scale (0 = no narrowing; 1 = up to 25% narrowing; 2 = 26-65% narrowing; 3 = 66-99% narrowing; and 4 = complete narrowing). Scores were summed to calculate the total score ranging from 0 (no narrowing) to 168 (maximum narrowing). A large increase in joint narrowing score is indicative of worsening, whereas a small change or no change is indicative of inhibition of JSN.
Time Frame: Baseline and Weeks 52 and 104
Population: Full analysis set. Missing values were imputed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
units on a scale
  Week 52 | 2.0 (6.3) | 1.3 (6.6) | 0.5 (4.2)
  Week 104 | 4.0 (10.9) | 2.6 (9.5) | 0.9 (5.1)

21. Secondary Outcome: Number of Participants With No Worsening in Modified Total Sharp Score or Components During the Double-blind Treatment Phase
Description: The number of participants with no worsening in the modified Total Sharp Score (mTSS) and in erosion and joint space narrowing (JSN) scores, where no worsening is defined as a change from Baseline of ≤ 0 in mTSS, erosion score and JSN score, at Weeks 52 and 104.
  Digitized images of radiographs of hands and feet obtained at screening and during the study were scored in a blinded manner. Joints were scored for erosions on a scale of 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale of 0 (no damage) to 4 (ankylosis or complete dislocation). Erosion scores and narrowing scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]). An increase in mTSS from Baseline represents disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease represents improvement.
Time Frame: Baseline and Weeks 52 and 104
Population: Full analysis set. Participants with missing data or who withdrew early were considered non-responders.
Measure: Number; unit: participants
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 257 | 274 | 268
participants
  Modified Total Sharp Score: Week 52 | 78 | 112 | 141
  Modified Total Sharp Score: Week 104 | 70 | 105 | 136
  Erosion Scoe: Week 52 | 91 | 133 | 158
  Erosion Score: Week 104 | 81 | 121 | 148
  Joint Space Narrowing Score: Week 52 | 127 | 159 | 190
  Joint Space Narrowing Score: Week 104 | 112 | 147 | 175

22. Secondary Outcome: Number of Participants With No Erosions at Baseline and No New Erosions at Weeks 52 and 104
Description: The number of participants with no erosions at Baseline and no erosions at Weeks 52 and 104, where no erosions and no new erosions are defined as an erosion score = 0.
  Digitized images of radiographs of hands and feet obtained at screening and during the study were scored in a blinded manner. Joints on each hand/wrist (17 joints) and each forefoot (6 joints) were scored for erosions on a scale of 0 = no erosions; 1 = 1 discrete erosion or ≤20% joint involvement; 2 = 2 separate quadrants with erosion or 21-40% joint involvement; 3 = 3 separate quadrants with erosion or 41-60% joint involvement; 4 = all 4 quadrants with erosion or 61-80% joint involvement; and 5 = extensive destruction with >80% joint involvement. Scores were summed to calculate the total erosion score, which ranges from 0 (no erosion) to 230 (worst).
Time Frame: Baseline and Weeks 52 and 104
Population: Full analysis set participants with no erosions at Baseline and non-missing data.
Measure: Number; unit: participants
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 11 | 16 | 20
participants
  Week 52 | 8 | 10 | 13
  Week 104 | 7 | 8 | 11

23. Secondary Outcome: Number of Participants With Non-Involved Joints at Baseline and No Newly Involved Joints at Weeks 52 and 104
Description: Number of participants with non-involved joints at Baseline and no newly involved joints at Weeks 52 and 104, where involved joints or no newly involved joints are defined as modified Total Sharp Score (mTSS) = 0.
  Digitized images of radiographs of hands and feet obtained at screening and during the study were scored in a blinded manner. Joints were scored for erosions on a scale of 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale of 0 (no damage) to 4 (ankylosis or complete dislocation). Erosion scores and narrowing scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]).
Time Frame: Baseline and Weeks 52 and 104
Population: Full analysis set participants with non-involved joints at Baseline and non-missing data.
Measure: Number; unit: participants
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 5 | 14 | 16
participants
  Week 52 | 4 | 9 | 12
  Week 104 | 3 | 7 | 9

24. Secondary Outcome: Number of Participants Meeting ACR20 Response Criteria Over 10 Years by Adalimumab Exposure
Description: American College of Rheumatology 20% (ACR20) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 20% improvement in tender joint count;
  * ≥ 20% improvement in swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * Acute phase reactant value (C-Reactive Protein).
  Baseline is the last value prior to the first dose of adalimumab. For participants randomized to the methotrexate (MTX) arm in the double-blind (DB) phase, Baseline was the last visit prior to the first adalimumab dose at Week 106 of the open-label (OL) phase.
Time Frame: Baseline and after 1, 2, 5, and 10 years of adalimumab exposure. Baseline was the last value prior to the first dose of adalimumab.
Population: Intent-to-treat (ITT) Analysis Set (all patients who received at least 1 dose of adalimumab during the study, including patients who received their first dose during the DB phase and those who received MTX during the DB phase and adalimumab in the OL phase) with available ACR data. "N" indicates patients with non-missing data at each time point.
Measure: Number; unit: participants
Groups:
- Any Adalimumab: Participants received either methotrexate (MTX), adalimumab, or methotrexate + adalimumab during the 2-year double-blind treatment phase. During the 8-year open-label phase all participants received adalimumab 40 mg every other week.
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 687
participants
  Year 1 [N=410] | 340
  Year 2 [N=385] | 332
  Year 5 [N=325] | 231
  Year 10 [N=170] | 154

25. Secondary Outcome: Number of Participants Meeting ACR50 Response Criteria Over 10 Years by Adalimumab Exposure
Description: American College of Rheumatology 50% (ACR50) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 50% improvement in tender joint count;
  * ≥ 50% improvement in swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * Acute phase reactant value (C-Reactive Protein).
  Baseline is the last value prior to the first dose of adalimumab. For patients randomized to the methotrexate (MTX) arm in the double-blind (DB) phase, Baseline was the last visit prior to the first adalimumab dose at Week 106 of the open-label (OL) phase.
Time Frame: as for outcome 24
Population: ITT Analysis Set with available ACR data. "N" indicates patients with non-missing data at each time point.
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 687
participants
  Year 1 [N=410] | 269
  Year 2 [N=385] | 266
  Year 5 [N=325] | 194
  Year 10 [N=170] | 127

26. Secondary Outcome: Number of Participants Meeting ACR70 Response Criteria Over 10 Years by Adalimumab Exposure
Description: American College of Rheumatology 70% (ACR70) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 70% improvement in tender joint count;
  * ≥ 70% improvement in swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * Acute phase reactant value (C-Reactive Protein).
  Baseline is the last value prior to the first dose of adalimumab. For patients randomized to the methotrexate (MTX) arm in the double-blind (DB) phase, Baseline was the last visit prior to the first adalimumab dose at Week 106 of the open-label (OL) phase.
Time Frame: as for outcome 24
Population: ITT Analysis Set with available data. "N" indicates patients with non-missing data at each time point.
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 687
participants
  Year 1 [N=410] | 186
  Year 2 [N=385] | 207
  Year 5 [N=325] | 153
  Year 10 [N=170] | 102

27. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire - Disability Index (HAQ-DI) Over 10 Years by Adalimumab Exposure
Description: as for outcome 3
Time Frame: Baseline and Years 1, 2, 5, and 10. Baseline was the last value prior to the first dose of adalimumab. For patients randomized to the MTX arm in the DB phase, Baseline was the last visit prior to the first adalimumab dose at Week 106.
Population: ITT Analysis Set, with available data. "N" indicates patients with non-missing data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 692
units on a scale
  Year 1 [N=407] | -0.9 (0.68)
  Year 2 [N=390] | -0.9 (0.70)
  Year 5 [N=344] | -0.7 (0.73)
  Year 10 [N=170] | -0.9 (0.73)

28. Secondary Outcome: Change From Baseline in DAS28 Over 10 Years by Adalimumab Exposure
Description: as for outcome 18
Time Frame: as for outcome 27
Population: ITT Analysis Set, with available data. "N" indicates patients with non-missing data at Baseline and the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 689
units on a scale
  Year 1 [N=403] | -3.2 (1.49)
  Year 2 [N=386] | -3.3 (1.61)
  Year 5 [N=330] | -2.8 (1.93)
  Year 10 [N=158] | -3.9 (1.29)

29. Secondary Outcome: Number of Participants With DAS28 < 2.6 and < 3.2 Over 10 Years by Adalimumab Exposure
Description: as for outcome 18
Time Frame: After 1, 2, 5, and 10 years of adalimumab exposure
Population: ITT Analysis Set, with available data. The Number of Participants Analyzed indicates patients with non-missing DAS28 scores at any post-baseline time point; "N" indicates patients with non-missing data at each specified time point.
Measure: Number; unit: participants
Groups:
- Adalimumab: DAS28 < 2.6: Participants with a DAS28 score less than 2.6, who received either methotrexate (MTX), adalimumab, or methotrexate + adalimumab during the 2-year double-blind treatment phase and adalimumab 40 mg every other week during the 8-year open-label phase.
- Adalimumab: DAS28 < 3.2: Participants with a DAS28 score less than 3.2, who received either methotrexate (MTX), adalimumab, or methotrexate + adalimumab during the 2-year double-blind treatment phase and adalimumab 40 mg every other week during the 8-year open-label phase.
Arm/Group | Adalimumab: DAS28 < 2.6 | Adalimumab: DAS28 < 3.2
Number analyzed (Participants) | 694 | 694
participants
  Year 1 [N=405] | 173 | 244
  Year 2 [N=389] | 215 | 271
  Year 5 [N=333] | 190 | 244
  Year 10 [N=159] | 109 | 135

30. Secondary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) Over 10 Years
Description: The modified TSS (mTSS) is a measure of change in joint health. Digitized images of radiographs of hands and feet obtained at screening and during the study were scored in a blinded manner. Joints were scored for erosions on a scale of 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale of 0 (no damage) to 4 (ankylosis or complete dislocation). Erosion scores and narrowing scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]). An increase in mTSS from Baseline represents disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease represents improvement.
Time Frame: Baseline (prior to first study drug treatment) and Years 2 and 10
Population: ITT Analysis Set, with available data. "N" indicates patients with non-missing radiographic data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 83 | 93 | 90
units on a scale
  Year 2 [N=83, 92, 89] | 6.3 (12.44) | 5.1 (9.63) | 0.3 (3.00)
  Year 10 [N= 83, 93, 90] | 10.8 (20.01) | 9.2 (15.21) | 3.9 (9.64)

31. Secondary Outcome: Number of Participants With No Radiographic Progression Over 10 Years
Description: The modified Total Sharp Score (mTSS) is a measure of change in joint health. Digitized images of radiographs of hands and feet obtained at screening and during the study were scored in a blinded manner. Joints were scored for erosions on a scale of 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale of 0 (no damage) to 4 (ankylosis or complete dislocation). Erosion scores and narrowing scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]). An increase in mTSS from Baseline represents disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease represents improvement. The number of participants with change from Baseline ≤ 0.5 and ≤ 0 is reported as a measure of no disease progression.
Time Frame: Baseline (prior to first study drug treatment) and Years 2 and 10.
Population: ITT Analysis Set, with available data. "N" indicates patients with non-missing radiographic data at each time point.
Measure: Number; unit: participants
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 83 | 93 | 90
participants
  Change ≤ 0.5 at Year 2 [N=83, 92, 89] | 36 | 40 | 65
  Change ≤ 0.5 at Year 10 [N=83, 93, 90] | 26 | 22 | 33
  Change ≤ 0 at Year 2 [N=83, 92, 89] | 22 | 30 | 51
  Change ≤ 0 at Year 10 [N=83, 93, 90] | 19 | 16 | 29

32. Secondary Outcome: Composite Score of ACR50 Plus No Change in Modified Total Sharp Score
Time Frame: Year 10
Population: This outcome measure was not analyzed due to a protocol amendment.
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate
Number analyzed (Participants) | 0 | 0 | 0

33. Secondary Outcome: Number of Participants With a Major Clinical Response Over 10 Years by Adalimumab Exposure
Description: A major clinical response was defined as maintenance of an ACR70 response for at least a 6-month continuous period at any time during the study following the first dose of adalimumab. A participant was a responder if the following criteria for improvement from Baseline were met:
  * ≥ 70% improvement in tender joint count;
  * ≥ 70% improvement in swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * Acute phase reactant value (C-Reactive Protein).
Time Frame: From the first dose of adalimumab (at Week 1 or Week 106 for patients initially randomized to methotrexate in the DB phase) to Year 10
Population: ITT Analysis Set for participants with non-missing ACR data.
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 687
participants | 273

34. Secondary Outcome: Number of Participants With Improvement in HAQ-DI by 0.22 and 0.5 Units Over 10 Years by Adalimumab Exposure
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. A decrease in the HAQ-DI score represents an improvement in physical function; a clinically significant improvement is defined as a decrease of least 0.22 from Baseline in the HAQ-DI score. The number of participants with improvement in HAQ-DI of at least 0.22 and 0.5 units from Baseline is reported.
Time Frame: as for outcome 27
Population: ITT Analysis Set, with available data. The Number of Participants Analyzed indicates patients with non-missing HAQ-DI scores at any post-baseline time point; "N" indicates patients with non-missing data at each specified time point.
Measure: Number; unit: participants
Groups:
- Adalimumab: HAQ Decrease ≥ 0.22: Participants with a decrease of least 0.22 in HAQ from baseline, who received either methotrexate (MTX), adalimumab, or methotrexate + adalimumab during the 2-year double-blind treatment phase and adalimumab 40 mg every other week during the 8-year open-label phase.
- Adalimumab: HAQ Decrease ≥ 0.5: Participants with a decrease of least 0.5 in HAQ from baseline, who received either methotrexate (MTX), adalimumab, or methotrexate + adalimumab during the 2-year double-blind treatment phase and adalimumab 40 mg every other week during the 8-year open-label phase.
Arm/Group | Adalimumab: HAQ Decrease ≥ 0.22 | Adalimumab: HAQ Decrease ≥ 0.5
Number analyzed (Participants) | 692 | 692
participants
  Year 1 [N=407] | 353 | 285
  Year 2 [N=390] | 324 | 265
  Year 5 [N=344] | 239 | 188
  Year 10 [N=170] | 140 | 112

ADVERSE EVENTS:
Time Frame: For the double-blind treatment phase, up to 2 years (Methotrexate, Adalimumab and Adalimumab + Methotrexate reporting groups). For the Any Adalimumab reporting group, adverse events include the open-label extension, and are reported for up to 10 years.
Groups:
- Any Adalimumab: Participants received either methotrexate, adalimumab, or methotrexate + adalimumab during the 2-year double-blind treatment phase. During the 8-year open-label phase all participants received adalimumab 40 mg every other week.
  Adverse events reported include those that occurred at any time during adalimumab exposure (up to 10 years).
Arm/Group | Methotrexate | Adalimumab | Adalimumab + Methotrexate | Any Adalimumab
Serious Adverse Events (participants affected / at risk) | 47/257 | 65/274 | 56/268 | 320/697
Other Adverse Events (participants affected / at risk) | 227/257 | 227/274 | 241/268 | 634/697
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=257) | Adalimumab (N=274) | Adalimumab + Methotrexate (N=268) | Any Adalimumab (N=697)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 6
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 2
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 2 | 0 | 3
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 8
Atrial Flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 2
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 3
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 2
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Mitral valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 7
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 2
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 1
Pleuropericarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 1
Sinoatrial block (Cardiac disorders) | 0 | 0 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1 | 2
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Otosclerosis (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Goitre (Endocrine disorders) | 1 | 0 | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 2
Blindness (Eye disorders) | 0 | 0 | 0 | 1
Blindness unilateral (Eye disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 2 | 0 | 3
Corneal disorder (Eye disorders) | 0 | 0 | 0 | 1
Corneal opacity (Eye disorders) | 0 | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 0 | 1
Necrotising scleritis (Eye disorders) | 1 | 0 | 0 | 0
Ocular hypertension (Eye disorders) | 1 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 4
Retinal disorder (Eye disorders) | 0 | 0 | 1 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 1 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal wall cyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 3
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Crohn's Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 1 | 3
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1
Calcinosis (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 5
Death (General disorders) | 0 | 1 | 0 | 1
Device dislocation (General disorders) | 0 | 0 | 0 | 1
Drug ineffective (General disorders) | 0 | 1 | 0 | 1
Dysplasia (General disorders) | 0 | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 0 | 1
Medical device complication (General disorders) | 0 | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 4
Oedema (General disorders) | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 0 | 3
Stent-graft endoleak (General disorders) | 0 | 0 | 0 | 1
Sudden cardiac death (General disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 3
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 3 | 8
Hepatic necrosis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1 | 1
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 2
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1
Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 1 | 1 | 4
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 2
Bartholin's abscess (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 4
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 4
Bursitis infective (Infections and infestations) | 0 | 1 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 2 | 4
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Corneal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Disseminated tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 3
Eczema infected (Infections and infestations) | 0 | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 1
Epstein-barr virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 3
Extradural abscess (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 3
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 0 | 1
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 1 | 1 | 5
Localised infection (Infections and infestations) | 0 | 0 | 0 | 3
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Meningitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 0 | 0 | 1 | 1
Mycobacterium marinum infection (Infections and infestations) | 0 | 0 | 0 | 1
Neurological infection (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1
Parotitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 15
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 3
Sepsis (Infections and infestations) | 0 | 0 | 0 | 4
Septic shock (Infections and infestations) | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1
Tuberculosis gastrointestinal (Infections and infestations) | 0 | 0 | 0 | 1
Tuberculous pleurisy (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 2
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 4
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 4
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post-operative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Testicular injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1
Blood culture positive (Investigations) | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0 | 1
CSF pressure increased (Investigations) | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 1
Heart rate increased (Investigations) | 0 | 0 | 0 | 1
Hepatitis c antibody positive (Investigations) | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 1 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 0 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 7
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 4
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4
Bone erosion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bone fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 8
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 7
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 23
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 6 | 16 | 3 | 38
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 3
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bladder cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 5
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lymphoma cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant melanoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 2
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 5
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 2
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 2
Cervical myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Clonus (Nervous system disorders) | 0 | 1 | 0 | 1
Dementia (Nervous system disorders) | 0 | 0 | 1 | 1
Dementia alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Hyperreflexia (Nervous system disorders) | 0 | 1 | 1 | 2
Intention tremor (Nervous system disorders) | 0 | 0 | 1 | 1
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 2 | 0 | 1 | 7
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 3
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 3
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 3
Depression suicidal (Psychiatric disorders) | 0 | 0 | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 6
Calculus Ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 2
Renal haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal mass (Renal and urinary disorders) | 0 | 0 | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 1 | 2
Dyspareunia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 2
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 1 | 1 | 4
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1 | 2
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 3
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Uterine cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 2
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 6
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Abortion induced (Surgical and medical procedures) | 0 | 0 | 0 | 1
Foot operation (Surgical and medical procedures) | 0 | 0 | 1 | 1
Female sterilization (Surgical and medical procedures) | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 2
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Aortitis (Vascular disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 4
Femoral artery occlusion (Vascular disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1
Iliac artery stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Rheumatoid vasculitis (Vascular disorders) | 0 | 1 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 1 | 2
Vasculitis (Vascular disorders) | 1 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=257) | Adalimumab (N=274) | Adalimumab + Methotrexate (N=268) | Any Adalimumab (N=697)
Anaemia (Blood and lymphatic system disorders) | 8 | 13 | 4 | 43
Lymphadenopathy (Blood and lymphatic system disorders) | 12 | 15 | 0 | 28
Vertigo (Ear and labyrinth disorders) | 9 | 14 | 5 | 42
Cataract (Eye disorders) | 5 | 5 | 6 | 39
Conjunctivitis (Eye disorders) | 3 | 6 | 10 | 36
Abdominal pain (Gastrointestinal disorders) | 9 | 11 | 12 | 46
Nausea (Gastrointestinal disorders) | 53 | 48 | 46 | 131
Dyspepsia (Gastrointestinal disorders) | 26 | 20 | 25 | 74
Diarrhoea (Gastrointestinal disorders) | 42 | 32 | 28 | 105
Abdominal pain upper (Gastrointestinal disorders) | 22 | 19 | 24 | 77
Vomiting (Gastrointestinal disorders) | 12 | 12 | 14 | 44
Mouth ulceration (Gastrointestinal disorders) | 15 | 7 | 12 | 25
Constipation (Gastrointestinal disorders) | 17 | 3 | 11 | 33
Chest pain (General disorders) | 8 | 13 | 12 | 42
Fatigue (General disorders) | 27 | 28 | 33 | 98
Oedema peripheral (General disorders) | 16 | 16 | 18 | 68
Pyrexia (General disorders) | 9 | 11 | 4 | 35
Nasopharyngitis (Infections and infestations) | 63 | 62 | 81 | 219
Gastroenteritis (Infections and infestations) | 11 | 6 | 9 | 38
Herpes zoster (Infections and infestations) | 2 | 8 | 4 | 50
Upper respiratory tract infection (Infections and infestations) | 47 | 24 | 50 | 176
Pharyngitis (Infections and infestations) | 11 | 9 | 10 | 43
Respiratory tract infection (Infections and infestations) | 3 | 10 | 8 | 38
Rhinitis (Infections and infestations) | 11 | 14 | 15 | 48
Sinusitis (Infections and infestations) | 17 | 23 | 29 | 111
Oral herpes (Infections and infestations) | 10 | 5 | 16 | 43
Urinary tract infection (Infections and infestations) | 22 | 30 | 21 | 132
Bronchitis (Infections and infestations) | 28 | 18 | 21 | 109
Influenza (Infections and infestations) | 18 | 21 | 15 | 77
Contusion (Injury, poisoning and procedural complications) | 8 | 5 | 19 | 48
Fall (Injury, poisoning and procedural complications) | 5 | 5 | 10 | 42
Alanine aminotransferase increased (Investigations) | 17 | 7 | 29 | 52
Aspartate aminotransferase increased (Investigations) | 11 | 4 | 14 | 28
Hypercholesterolaemia (Metabolism and nutrition disorders) | 8 | 12 | 2 | 61
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 34 | 30 | 129
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 31 | 23 | 108
Bursitis (Musculoskeletal and connective tissue disorders) | 6 | 11 | 10 | 58
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 9 | 12 | 40
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 9 | 5 | 46
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 6 | 4 | 39
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 9 | 2 | 50
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 11 | 18 | 74
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 38 | 43 | 26 | 189
Joint swelling (Musculoskeletal and connective tissue disorders) | 13 | 15 | 5 | 39
Tendonitis (Musculoskeletal and connective tissue disorders) | 5 | 5 | 5 | 41
Headache (Nervous system disorders) | 42 | 59 | 55 | 155
Dizziness (Nervous system disorders) | 15 | 26 | 20 | 67
Paraesthesia (Nervous system disorders) | 8 | 13 | 8 | 46
Depression (Psychiatric disorders) | 19 | 13 | 19 | 69
Insomnia (Psychiatric disorders) | 7 | 17 | 8 | 48
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 34 | 30 | 107
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 16 | 10 | 43
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 | 24 | 22 | 65
Alopecia (Skin and subcutaneous tissue disorders) | 13 | 11 | 18 | 38
Rash (Skin and subcutaneous tissue disorders) | 22 | 25 | 17 | 98
Eczema (Skin and subcutaneous tissue disorders) | 6 | 12 | 9 | 43
Erythema (Skin and subcutaneous tissue disorders) | 3 | 9 | 5 | 36
Hypertension (Vascular disorders) | 32 | 25 | 29 | 153
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 9 | 8 | 48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.